CLINICAL TRIAL: NCT01309087
Title: Airway Epithelium Gene Expression in the Diagnosis of Lung Cancer: AEGIS CLIA
Acronym: AEGIS
Status: Completed | Type: Observational
Sponsor: Allegro Diagnostics, Corp. (Industry)
Collaborators: Beth Israel Deaconess Medical Center (Other); Columbia University (Other); Vanderbilt University (Other); University of British Columbia (Other); University of Pennsylvania (Other); New York University (Other); Temple University (Other); Indiana University (Other); University of Alabama at Birmingham (Other); University of Virginia (Other); University of Missouri-Columbia (Other); Louisiana State University Health Sciences Center in New Orleans (Other); University of Dublin, Trinity College (Other); Georgia Lung Associates PC (Other)
Responsible Party: Sponsor
Other Study IDs: ADx-0001: AEGIS CLIA
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Lung Cancer
Keywords: Gene Expression; Lung Cancer; Smoking
MeSH Terms: conditions — Lung Neoplasms; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cells, Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to substantiate prediction accuracy(with a tighter 95% confidence interval compared to current diagnostic modalities), of a lung cancer biomarker for risk stratification of patients into high and low risk categories to aid in clinical evaluation of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is being evaluated for the diagnosis of possible lung cancer or "rule out lung cancer" and is indicated for bronchoscopy.
2. The patient is undergoing bronchoscopy
3. ≥ 21 years of age
4. Patient meets local site's standard of care (SOC) for performing diagnostic bronchoscopy
5. The patient is a current or former cigarette smoker (defined as having smoked >100 cigarettes in their lifetime.

Exclusion Criteria:

1. The Pulmonary physician does not recommend that bronchoscopy be performed
2. The patient is unable to be consented into the study or unable to comply with requirements of the study
3. The patient has previously been diagnosed with primary lung cancer
4. Immediately prior to bronchoscopy, the patient has been on a mechanical ventilator for ≥ 24 consecutive hours.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are undergoing clinically indicated bronchoscopy for rule out lung cancre and have a history of cigarette smoking
Sampling Method: Non-Probability Sample
Enrollment: 756 (Actual)
Dates: Start 2009-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Primary Lung Cancer | One year from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Duncan Whitney, PhD, Study Director — Allegro Diagnostics
Locations (14):
- United States (12):
  - University of Alabama, Birmingham, Alabama
  - Georgia Lung Associates, Austell, Georgia
  - Indiana University, Indianapolis, Indiana
  - LSU, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Missouri, Columbia, Missouri
  - New York University, New York, New York
  - Columbia University, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia
- University of British Columbia, Vancouver, British Columbia, Canada
- Trinity College, Dublin, Ireland

REFERENCES:
- [Derived] Vachani A, Whitney DH, Parsons EC, Lenburg M, Ferguson JS, Silvestri GA, Spira A. Clinical Utility of a Bronchial Genomic Classifier in Patients With Suspected Lung Cancer. Chest. 2016 Jul;150(1):210-8. doi: 10.1016/j.chest.2016.02.636. Epub 2016 Feb 16. PMID 26896702
- [Derived] Silvestri GA, Vachani A, Whitney D, Elashoff M, Porta Smith K, Ferguson JS, Parsons E, Mitra N, Brody J, Lenburg ME, Spira A; AEGIS Study Team. A Bronchial Genomic Classifier for the Diagnostic Evaluation of Lung Cancer. N Engl J Med. 2015 Jul 16;373(3):243-51. doi: 10.1056/NEJMoa1504601. Epub 2015 May 17. PMID 25981554